CLINICAL TRIAL: NCT03491098
Title: The Efficacy of Nasal Steroids in Treatment of Otitis Media With Effusion: Acomparative Study
Acronym: Efficacy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muteea Mubark Salmen Bakuwiri (Other)
Responsible Party: Sponsor-Investigator, Muteea Mubark Salmen Bakuwiri, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Efficacy of Nasal Steroids
Record Dates: First submitted 2018-03-24; First posted 2018-04-09 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Otitis Media With Effusion
Keywords: Otitis Media with Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — prednisolone phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- momestone furoate spray first group: will be given (Placebo Comparator): Nasonex spray one puff in each nostril daily for 8 weeks
  Interventions: Drug: Mometasone Furoate spray
- prednisolone sodium phosphate 15mg second group: will be given (Placebo Comparator): Predsol fort tablet three times per day for 1 week then gradual withdrawal over 2 weeks
  Interventions: Drug: prednisolone sodium phosphate 15mg
- hypertonic sea water solution spray third group: will be given (Placebo Comparator): Nasal spray one puff in each nostril daily for 8 weeks
  Interventions: Drug: hypertonic sea water solution spray

INTERVENTIONS:
Drug: Mometasone Furoate spray — Mometasone Furoate spray one puff in each nostril daily for 8 weeks
  hypertonic sea water solution spray one puff in each nostril daily for (8) weeks.
  Arms: momestone furoate spray first group: will be given
Drug: prednisolone sodium phosphate 15mg — three times per day for 1 week then gradual withdrawal over 2 weeks
  Arms: prednisolone sodium phosphate 15mg second group: will be given
Drug: hypertonic sea water solution spray — one puff in each nostril daily for 8 weeks
  Arms: hypertonic sea water solution spray third group: will be given

SUMMARY:
Otitis media with effusion (OME) is defined as effusion in the middle ear without signs and symptoms of an acute infection. It is a leading cause of hearing impairment in children, and its early and proper management can avoid hearing and speech impairment, which can cause developmental delay in children.Although many conditions such as enlarged adenoids, cleft palate, Down syndrome, Kartagener syndrome, and nasopharyngeal neoplasm are related to the role of eustachian tube (ET) dysfunction in the pathogenesis of OME, allergic, immunologic, and infectious factors have also been claimed. Treatment of OME is still a controversial issue, as conventional treatment approaches fail to provide satisfactory and permanent relief of otologic symptoms.There is lack of proven effectiveness of the commonly given treatments, such as antibiotics, decongestants, and antihistamines, which are potentially harmful and have disadvantages. Few in those studies,investigated topical intranasal steroid for OME treatment,and in those studies, the duration of intranasal steroid application was short and there was no hearing evaluation.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy of nasal steroids in management of OME by comparing its results with that of oral steroids and that of nasal saline spray.

Sixty patients (4-12) years aged children with OME over a period for two months will be included in this study. Informed written consent will obtained from the parents of patient studied after explanation of the research purpose.

Patient diagnosed clinically to have OME with type B tympanogram and conductive hearing loss will be enrolled in our study.

Exclusion criteria:

1. Patients previously managed by ventilation tube.
2. Those who had cleft palate. The patients were divided into three equal groups. In group 1, 20 patients will be received steroids spray, for. 2 months In group 2, 20 patients will be received steroids for 1 month In group 3, 20 patients will be receive hypertonic sea water solution Otoscopic examination, basic audiological evaluation including pure tone audiometry, and immittancemetry will be performed before treatment and repeated at 3 and 6 months after treatment. The evaluation was performed using ORBITR 922 VERSION2 . Examiners will be blinded to the type of treatment.

Tympanometry results were distinguished into four grades as classified by El-Anwar et al12: type A, normal curve (pressure 50/_99 H2O); type C1 (negative pressure _100/_199 mm H2O); type C2 (negative pressure _200/_394 mm H2O); type B (flat curve).2,3,11 The average hearing thresholds at 500 Hz and 1, 2, and 4 kHz were used in the statistical comparison.

Follow-up clinical examinations were done once per week for 3 weeks, at the end of treatment. The efficacy of nasal steroid for management of OME was compared with that of oral steroid and that of nasal sinomarin spray as placebo.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients (4-12) years aged children with OME over a period for two months.

Exclusion Criteria:

* Patients previously managed by ventilation tube.
* Those who had cleft palate.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical examination:Hearing loss | 2 weeks evaluation for 2 months
  Hearing loss,0=no symptoms,1= present 2 weeks ,3=present daily,4=always present,
Clinical examination:Nasal obstruction | 2 weeks evaluation for 2 months
  Nasal obstruction,0=no symptoms,1= present 2 weeks ,3=present daily,4=always present,
Full E.N.T history | 2 weeks evaluation for 2 months
  Snoring ,sleep apnea ,difficult suckling in infants,anterior nasal discharge and conductive hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Ezzat M Saleh, Professor, Study Chair — Assiut University; Mohamed M Abd ElNaeem, doctor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yousaf M, Inayatullah, Khan F. Medical versus surgical management of otitis media with effusion in children. J Ayub Med Coll Abbottabad. 2012 Jan-Mar;24(1):83-5. PMID 23855103
- [Background] Bernstein JM, Lee J, Conboy K, Ellis E, Li P. Further observations on the role of IgE-mediated hypersensitivity in recurrent otitis media with effusion. Otolaryngol Head Neck Surg. 1985 Oct;93(5):611-5. doi: 10.1177/019459988509300508. PMID 3932928
- [Background] Tomonaga K, Kurono Y, Chaen T, Mogi G. Adenoids and otitis media with effusion: nasopharyngeal flora. Am J Otolaryngol. 1989 May-Jun;10(3):204-7. doi: 10.1016/0196-0709(89)90064-1. PMID 2500860
- [Background] Ho WK, Wei WI, Yuen AP, Hui Y, Wong SH. Otorrhea after grommet insertion for middle ear effusion in patients with nasopharyngeal carcinoma. Am J Otolaryngol. 1999 Jan-Feb;20(1):12-5. doi: 10.1016/s0196-0709(99)90045-5. PMID 9950108
- [Background] Tang NL, Choy AT, John DG, van Hasselt CA. The otological status of patients with nasopharyngeal carcinoma after megavoltage radiotherapy. J Laryngol Otol. 1992 Dec;106(12):1055-8. doi: 10.1017/s0022215100121747. PMID 1487659